CLINICAL TRIAL: NCT05143606
Title: Fiberoptic Intubation Skill Performance After Self-directed Training Among Anesthesiology Residents: A Randomized Comparison of a 3D-printed Model Simulator and a Virtual Reality Software
Brief Title: 3D Printed Model Simulator or Virtual Reality Software for Training Fiberoptic Intubation Skill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Panop Limratana, Lecturer, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 877/2021
Record Dates: First submitted 2021-11-18; First posted 2021-12-03 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Intubation, Endotracheal
Keywords: Fiberoptic bronchoscopy; intubation skill; deliberate practice

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors are blinded to each participant's group allocation. The assessors will be provided with video clips of the participants performing FOI. The identity and group allocation of each participant will not be revealed during the assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printed simulator (Experimental): The participants in this arm will undergo two self-directed training sessions on a custom-made 3D-printed airway simulator. The participants will use a standard intubating fiberoptic bronchoscope to practice fiberoptic-assisted nasal intubation.
  The sessions will be one week apart. Each session is 30 minutes per participant.
  Interventions: Other: 3D-printed airway simulator
- Virtual reality software (Experimental): The participants in this arm will practice fiberoptic-assisted nasal intubation using the free virtual reality software (AirwayEX) on their mobile phones or computer tablets. Two practice sessions are required by the investigators. The sessions will be one week apart. Each session is 30 minutes per participant.
  The participants in this arm will have the opportunity to practice on the software as often as they feel necessary. All the additional practice data will be recorded.
  Interventions: Other: virtual reality software, AirwayEx

INTERVENTIONS:
Other: 3D-printed airway simulator — Two self-directed training on a standard fiberoptic bronchoscope and a custom-made 3D airway simulator.
  Arms: 3D printed simulator
Other: virtual reality software, AirwayEx — Two self-directed training on AirwayEx. With additional training as necessary.
  Arms: Virtual reality software

SUMMARY:
Fiberoptic-assisted intubation is an advanced skill that requires learners' practice as well as clinical experience during the anesthesiology residency training period. Current training methods including airway simulators and virtual reality software are used by medical schools worldwide.

The objective of this study is to compare the learner's fiberoptic intubation performance between training with a 3D-printed simulator and a virtual reality software.

DETAILED DESCRIPTION:
Fiberoptic-assisted intubation (FOI) is an essential skill of an anesthesiologist. It requires comprehensive knowledge of the airway anatomy and the proper and skillful use of a fiberoptic bronchoscope.

Fiberoptic-assisted intubations are usually performed in emergency situations and during difficult airway patient encounters. These situations are not ideal for learners to properly practice the skill.

The process of acquiring FOI skills includes teaching by experienced instructors, self-practice using commercially-available airway simulators, and practicing on virtual reality software.

The airway simulators and virtual reality software have their advantages and disadvantages.

In this randomized study, the investigators will compare the fiberoptic intubation skill among anesthesiology residents after self-training on a custom-made 3D simulator and self-training on a virtual reality software.

ELIGIBILITY:
Inclusion Criteria:

* Second-year anesthesiology resident

Exclusion Criteria:

* Refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Global rating scale score for fiberoptic intubation performance (GRS scale) | 1 week after self-directed practice session
  The 5-point rating scale assessing multiple aspects of fiberoptic intubation performance.
  The assessment includes, on the scale of 1 (minimum score) to 5 (maximum score), the following;
  1. Control
  2. Progression
  3. Orientation
  4. Views and collision
  5. Accuracy

SECONDARY OUTCOMES:
Time to successful intubation | 1 week after self-directed practice session
  The duration measured from the passing of the fiberoptic bronchoscope through the nasal opening and the time of successful intubation (defined as the passing of the endotracheal tube into the trachea above the carina).
  The measured duration is reported as seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apfelbaum JL, Hagberg CA, Caplan RA, Blitt CD, Connis RT, Nickinovich DG, Hagberg CA, Caplan RA, Benumof JL, Berry FA, Blitt CD, Bode RH, Cheney FW, Connis RT, Guidry OF, Nickinovich DG, Ovassapian A; American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Practice guidelines for management of the difficult airway: an updated report by the American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Anesthesiology. 2013 Feb;118(2):251-70. doi: 10.1097/ALN.0b013e31827773b2. No abstract available. PMID 23364566
- [Background] Wiles MD, McCahon RA, Armstrong JAM. An Audit of Fibreoptic Intubation Training Opportunities in a UK Teaching Hospital. Journal of Anesthesiology. 2014;703820.
- [Background] Clarke RC, Gardner AI. Anaesthesia trainees' exposure to airway management in an Australian tertiary adult teaching hospital. Anaesth Intensive Care. 2008 Jul;36(4):513-5. PMID 18714618
- [Background] Naik VN, Matsumoto ED, Houston PL, Hamstra SJ, Yeung RY, Mallon JS, Martire TM. Fiberoptic orotracheal intubation on anesthetized patients: do manipulation skills learned on a simple model transfer into the operating room? Anesthesiology. 2001 Aug;95(2):343-8. doi: 10.1097/00000542-200108000-00014. PMID 11506104
- [Background] Chao I, Young J, Coles-Black J, Chuen J, Weinberg L, Rachbuch C. The application of three-dimensional printing technology in anaesthesia: a systematic review. Anaesthesia. 2017 May;72(5):641-650. doi: 10.1111/anae.13812. Epub 2017 Jan 27. PMID 28127746
- [Background] Carter JC, Broadbent J, Murphy EC, Guy B, Baguley KE, Young J. A three-dimensional (3D) printed paediatric trachea for airway management training. Anaesth Intensive Care. 2020 May;48(3):243-245. doi: 10.1177/0310057X20925827. Epub 2020 Jun 14. PMID 32536185
- [Background] Jiang B, Ju H, Zhao Y, Yao L, Feng Y. Comparison of the Efficacy and Efficiency of the Use of Virtual Reality Simulation With High-Fidelity Mannequins for Simulation-Based Training of Fiberoptic Bronchoscope Manipulation. Simul Healthc. 2018 Apr;13(2):83-87. doi: 10.1097/SIH.0000000000000299. PMID 29621098
- [Background] Giglioli S, Boet S, De Gaudio AR, Linden M, Schaeffer R, Bould MD, Diemunsch P. Self-directed deliberate practice with virtual fiberoptic intubation improves initial skills for anesthesia residents. Minerva Anestesiol. 2012 Apr;78(4):456-61. Epub 2012 Feb 6. PMID 22310190
- [Background] Kadys A, Rancevienė D, Macas A. Using Smartphone Application iLarynx to Teach Novices to Perform Fiber Optic Intubation. Nursing education, research, & practice: NERP. Kaunas: Lietuvos sveikatos mokslų universitetas, 2016, vol. 6, no. 1. 2016.
- [Background] Ho BHK, Chen CJ, Tan GJS, Yeong WY, Tan HKJ, Lim AYH, Ferenczi MA, Mogali SR. Multi-material three dimensional printed models for simulation of bronchoscopy. BMC Med Educ. 2019 Jun 27;19(1):236. doi: 10.1186/s12909-019-1677-9. PMID 31248397
- [Background] Chan JK, Ng I, Ang JP, Koh SM, Lee K, Mezzavia P, Morris J, Loh F, Segal R. Randomised controlled trial comparing the Ambu(R) aScope2 with a conventional fibreoptic bronchoscope in orotracheal intubation of anaesthetised adult patients. Anaesth Intensive Care. 2015 Jul;43(4):479-84. doi: 10.1177/0310057X1504300410. PMID 26099760
- [Background] K Latif R, Bautista A, Duan X, Neamtu A, Wu D, Wadhwa A, Akca O. Teaching basic fiberoptic intubation skills in a simulator: initial learning and skills decay. J Anesth. 2016 Feb;30(1):12-9. doi: 10.1007/s00540-015-2091-z. Epub 2015 Oct 22. PMID 26493397